CLINICAL TRIAL: NCT04995484
Title: An Open-Label, Single-Dose Study to Investigate the Influence of Hepatic Impairment on the Pharmacokinetics of MK-6482
Brief Title: A Study of Belzutifan (MK-6482) in Participants With Hepatic Impairment (MK-6482-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-020; MK-6482-020 (Other: Merck)
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Moderate Hepatic Impairment
MeSH Terms: interventions — belzutifan

STUDY DESIGN:
Intervention Model Description: Parallel Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment will receive a single oral 80 mg dose of belzutifan on Day 1.
  Interventions: Drug: Belzutifan
- Healthy (Experimental): Participants with normal hepatic function will receive a single oral 80 mg dose of belzutifan on Day 1.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Two 40 mg tablets given as a single oral 80 mg dose.
  Other Names: MK-6482; PT2977; WELIREG

SUMMARY:
The primary purpose of this study is to compare the plasma pharmacokinetics (PK) of belzutifan (MK-6482) following a single oral 80 mg dose of belzutifan in participants with moderate hepatic impairment to that of healthy matched control participants. This study will also evaluate the safety and tolerability of a single oral 80 mg dose of belzutifan in participants with moderate hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* Is in good health.
* Has a body mass index (BMI) 18.0-40.0 kg/m^2.

For Participants With Normal Hepatic Function:

Male Participants -Must have been vasectomized or surgically sterilized for at least 4 months or more prior to study intervention administration and agree to the following during the intervention period and for at least 5 days after administration of study intervention, be abstinent from heterosexual intercourse as their preferred and usual lifestyle or must agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a woman of childbearing potential (WOCBP) who is not currently pregnant.

Female Participants

-Is a woman of non-childbearing potential (WONCBP).

For Participants With Moderate Hepatic Impairment

* Has a diagnosis of chronic (>6 months), stable (no acute episodes of illness within the previous 30 days from administration of study intervention due to deterioration in hepatic function) hepatic impairment.
* Has a score on the Child-Pugh scale of B (a score of 7-9 on Child-Pugh Score)

Male Participants -Have been vasectomized or surgically sterilized for at least 4 months or more prior to study intervention administration and agree to the following during the intervention period and for at least 5 days after administration of study intervention, be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent or must agree to use a male condom plus partner use of an additional contraceptive method when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.

Female Participants

- Must be a WONCBP.

Exclusion Criteria:

All Participants:

* Is a heavy smoker or heavy user of nicotine-containing products (>20 cigarettes or equivalent/day).
* Consumes greater than 3 glasses of alcoholic beverages or equivalent per day.
* Consumes excessive amounts, defined as greater than 6 servings of caffeinated beverages per day.
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within the last 2 years.
* Presents any concern by the investigator regarding safe participation in the study.

For Participants with Normal Hepatic Function

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Is mentally or legally incapacitated, has significant emotional problems or has a history of clinically significant psychiatric disorder of the last 5 years.
* Has a history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood within the last 4 weeks.
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs (with the exception of prescription drugs that are approved by the investigator and Sponsor) or herbal remedies for the prohibited period of time.
* Has received any nonlive vaccine starting from 14 days prior to study intervention or is scheduled to receive any nonlive vaccine through 30 days following study intervention. Exception: COVID-19 vaccine may be administered.
* Has participated in another investigational study within 4 weeks prior to study intervention administration.

For Participants With Moderate Hepatic Impairment

* Is mentally or legally incapacitated, has significant emotional problems or has a history of clinically significant psychiatric disorder in the last 5 years.
* Has a history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
* Has fluctuating or rapidly deteriorating hepatic function.
* Has a history of liver or other solid organ transplantation.
* Has transjugular intrahepatic portosystemic shunt and/or has undergone portacaval shunting.
* Has encephalopathy Grade 3 or worse within 28 days before administration of study intervention.
* Is positive for HIV.
* Has had major surgery, donated or lost 1 unit of blood within the last 4 weeks.
* Is unable to refrain from or anticipates the use of any medication, including prescription and nonprescription drugs (with the exception of prescription drugs that are approved by the investigator and Sponsor) or herbal remedies for the prohibited period of time.
* Has received any nonlive vaccine starting from 14 days prior to study intervention or is scheduled to receive any nonlive vaccine through 30 days following study intervention. Exception: COVID-19 vaccine may be administered.
* Has participated in another investigational study within 4 weeks prior to study intervention administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Orlando Clinical Research Center ( Site 0001), Orlando, Florida
  - The Texas Liver Institute ( Site 0002), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single oral 80 mg dose of belzutifan on Day 1.
- Healthy: Participants with normal hepatic function received a single oral 80 mg dose of belzutifan on Day 1.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment | Healthy
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment | Healthy | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (2.69) | 61.4 (5.63) | 61.0 (4.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-Inf) of Belzutifan
Description: AUC0-Inf was defined as the area under the concentration-time curve of belzutifan from time zero to infinity. Blood samples collected predose and at multiple timepoints postdose were used to determine AUC0-Inf of belzutifan.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 72, 96, and 120 hours postdose
Population: All participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, who have available measurement data, and have no important protocol deviations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
ng*hr/mL | 22500 (80.3) | 14800 (35.1)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy; Test type: Other; Geometric Mean Ratio = 1.52, 90% CI 2-sided [0.95 to 2.43] — Moderate Hepatic Impairment/Healthy

2. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24hrs) of Belzutifan
Description: AUC0-24hrs was defined as the area under the concentration-time curve of belzutifan from time zero to 24 hours postdose. Blood samples collected predose and at multiple timepoints postdose were used to determine AUC0 to 24 hours of belzutifan.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
ng*hr/mL | 10500 (34.5) | 9650 (28.8)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy; Test type: Other; Geometric Mean Ratio = 1.09, 90% CI 2-sided [0.84 to 1.42] — Moderate Hepatic Impairment/Healthy

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Belzutifan
Description: Cmax was defined as the peak level belzutifan reaches in the blood. Blood samples collected predose and at multiple timepoints postdose were used to determine Cmax of belzutifan.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
ng/mL | 852 (28.7) | 870 (31.4)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy; Test type: Other; Geometric Mean Ratio = 0.98, 90% CI 2-sided [0.76 to 1.26] — Moderate Hepatic Impairment/Healthy

4. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Belzutifan
Description: Tmax was defined as the time it took belzutifan to reach its peak level in the blood. Blood samples collected predose and at multiple timepoints postdose were used to determine the Tmax of belzutifan.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
hr | 2.00 [0.50 to 3.00] | 2.00 [1.00 to 3.00]

5. Primary Outcome: Apparent Terminal Half-life (t1/2) of Belzutifan
Description: Apparent terminal half-life (t1/2) was defined as the time needed to reduce the level of belzutifan in the blood by one-half (1/2). Blood samples collected predose and at multiple timepoints postdose were used to determine the apparent terminal half-life (t1/2) of belzutifan.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 9, 12, 24, 36, 48, 72, 96, and 120 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
hr | 23.5 (70.5) | 15.4 (16.4)

6. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is reported.
Time Frame: Up to 15 days
Population: All participants who were allocated and received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
Participants | 1 | 1

7. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued the study due to an AE is reported.
Time Frame: Up to 15 days
Population: All participants who were allocated and received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hepatic Impairment | Healthy
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 days
Description: All Cause Mortality is reported for all allocated participants. Serious Adverse Events and Other Adverse Events are reported for all participants who received treatment.
Groups:
- Healthy Matched Control: Participants with normal hepatic function received a single oral 80 mg dose of belzutifan on Day 1.
Arm/Group | Moderate Hepatic Impairment | Healthy Matched Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 1/9 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hepatic Impairment (N=9) | Healthy Matched Control (N=8)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. A coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT04995484/Prot_SAP_000.pdf